CLINICAL TRIAL: NCT04891458
Title: Effect of Intraoperative Sedation on Perioperative Neurocognitive Disorders in Elderly Patients
Brief Title: Effect of Intraoperative Sedation on PND in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOSPND
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Elderly; Anesthesia
Keywords: Anesthesia; Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Anesthesiologists who provide anesthesia for patients need to adjust the dose of sedative drugs according to the score of MOAA/S during operation, so blind method is not used for anesthesiologists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients received lighter sedation with propofol after spinal anesthesia (Experimental): Continuous infusion of propofol at a rate of 1.0-4.0mg/kg per hour until the end of surgery to achieve MOAA/S 0-2.
  Interventions: Drug: Patients received lighter sedation with propofol after spinal anesthesia.
- Patients received heavier sedation with propofol after spinal anesthesia (Experimental): Continuous infusion of propofol at a rate of 1.0-4.0mg/kg per hour until the end of surgery to achieve MOAA/S 3-5.
  Interventions: Drug: Patients received heavier sedation with propofol after spinal anesthesia
- Patients received lighter sedation with dexmedetomidine after spinal anesthesia. (Experimental): Continuous infusion of dexmedetomidine at a rate of 0.2-0.7 mcg/ kg per hour until the end of surgery to achieve MOAA/S 0-2.
  Interventions: Drug: Patients received lighter sedation with dexmedetomidine after spinal anesthesia
- Patients received heavier sedation with dexmedetomidine after spinal anesthesia. (Experimental): Continuous infusion of dexmedetomidine at a rate of 0.2-0.7 mcg/ kg per hour until the end of surgery to achieve MOAA/S 3-5.
  Interventions: Drug: Patients received heavier sedation with dexmedetomidine after spinal anesthesia.

INTERVENTIONS:
Drug: Patients received lighter sedation with propofol after spinal anesthesia. — MOAA/S 0-2.
  Arms: Patients received lighter sedation with propofol after spinal anesthesia
Drug: Patients received heavier sedation with propofol after spinal anesthesia — MOAA/S 3-5.
  Arms: Patients received heavier sedation with propofol after spinal anesthesia
Drug: Patients received lighter sedation with dexmedetomidine after spinal anesthesia — MOAA/S 0-2.
  Arms: Patients received lighter sedation with dexmedetomidine after spinal anesthesia.
Drug: Patients received heavier sedation with dexmedetomidine after spinal anesthesia. — MOAA/S 3-5.
  Arms: Patients received heavier sedation with dexmedetomidine after spinal anesthesia.

SUMMARY:
The aim of this study was to identify the effects of different depths of sedation and choices of sedative drugs on perioperative neurocognitive disorders in the elderly patients receiving hip surgery under spinal anesthesia.

DETAILED DESCRIPTION:
PND is a complication of the central nervous system after anesthesia and surgery which is considered to be a common complication in elderly patients. Age is an independent risk factor for the occurrence of PND. Prolonged hospitalization, incapacity and long duration of PND aggravate the economic burden of individuals, families and society. The pathogenesis of PND is still unclear. Recent studies suggest that the blood-brain barrier (BBB) is damaged by surgery or anesthesia, which causes the activation of inflammatory factors such as TNF α and NF - κ B, and then leads to the decline of hippocampus cognitive function. In recent years, it has been found that dexmedetomidine can reduce the brain injury during ischemia-reperfusion and reduce the occurrence of PND. BDNF is a neurotrophin, which plays an important role in the growth, differentiation, synaptic plasticity, survival and repair of neurons. Studies have shown that the decrease of BDNF concentration is related to PND, which can be used as an index to evaluate brain injury and predict PND. S100 β protein is a specific low molecular calcium binding protein of nervous system which can be increased early after brain injury, so it can be used to reflect the severity and prognosis of brain injury and predict PND.In this randomized controlled trial, investigators will compare the incidence of PND in hip surgery with four intraoperative sedation regimens. After spinal anesthesia, the following sedation regimen will be used: (1) Intravenous infusion of propofol to make patients receive lighter sedation(modified observer's assessment of alertness/sedation score[MOAA/S],0-2) (2) Intravenous infusion of propofol to make patients receive heavier sedation(MOAA/S,3-5) (3)After a bolus of dexmedetomidine, intravenous infusion of dexmedetomidine to make patients receive lighter sedation(MOAA/S,0-2) (4) After a bolus of dexmedetomidine, intravenous infusion of dexmedetomidine to make patients receive heavier sedation(MOAA/S,3-5). 3ml venous blood samples were collected before anesthesia (T0), 1 h after operation (T1), 1 day after operation (T2) and 7 days after operation (T3). Plasma samples were collected after centrifugation and the concentrations of BDNF and S100 β were determined by ELISA. After 7days of surgery, PND is screened by CAM with a trained research assistant everyday, and CAM positive patients are judged by a qualified psychiatrist to meet DSM-V criteria until the patient is discharged. For patients with PND, the delirium rating scale (DRS) was used to assess the degree of delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Acquisition of informed consent,
2. Patients with hip fracture surgery under spinal anesthesia,
3. Grade I to III based on American Society of Anesthesiologists ASA classification,
4. Age ≥65.

Exclusion Criteria:

1. There was a history of cardiovascular and cerebrovascular adverse events in the past six months, including myocardial infarction, angina pectoris, severe arrhythmia, stroke or transient ischemic attack (TIA)
2. Heart failure (NYHA III / IV and / or LVEF < 30%)
3. Bradycardia
4. Respiratory failure (need oxygen)
5. Glasgow Coma Scale ≤ 14 points
6. Severe hepatic and renal insufficiency (child Pugh grade B or C)
7. Preoperative cognitive impairment or sedative drugs (benzodiazepines, etc.).
8. Adverse reactions such as allergy to dexmedetomidine or / or propofol
9. Preoperative bilateral hip fracture or other trauma need simultaneous operation
10. Contraindications of spinal anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | 1 week
  Postoperative delirium is assessed with the Confusion Assessment Method and in accordance with the the Diagnostic and Statistical Manual of Mental Disorders, 5th edition diagnostic criteria for delirium，each postoperative day until discharge.
  Delirium severity is scored using the long Confusion Assessment Method Severity score.
Change from Cognitive state in 1 week. | 1 week
  Cognitive state is measured with the Beijing version of Montreal Cognitive Assessment preoperatively，on the first day and the seventh day after surgery. A score of ≥26 is considered normal in Montreal Cognitive Assessment，with the maximum score of 30 points. The lower the score, the worse the cognitive status.

SECONDARY OUTCOMES:
Inflammatory biomarker level in blood | before anesthesia (T0), 1 hour after operation (T1), 1 day after operation (T2) and 7 days after operation (T3)
  BDNF、S100 β 、NF-κB、TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Zhao, PhD, Study Chair — Third Hospital of Hebei Medical University Department of Anesthesiology; Shuxing Zhu, M.D, Study Director — Third Hospital of Hebei Medical University Department of Anesthesiology; Xiuli Wang, PhD, Principal Investigator — Third Hospital of Hebei Medical University Department of Anesthesiology